CLINICAL TRIAL: NCT02018458
Title: Pilot Safety Trial of Preoperative Chemotherapy Combined With Dendritic Cell Vaccine in Patients With Locally Advanced, Triple-Negative Breast Cancer or ER-Positive, Her2-Negative Breast Cancer
Brief Title: Safety Study Of Chemotherapy Combined With Dendritic Cell Vaccine to Treat Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 013-154
Record Dates: First submitted 2013-12-04; First posted 2013-12-23 (Estimated); Results first posted 2020-03-13 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Dendritic cell vaccine; Breast Cancer; Doxorubicin; Paclitaxel; Cyclophosphamide; Carboplatin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LA TNBC: DC vaccine+Preop chemo (Experimental): LA TNBC patients will receive standard preop AC followed by TCb chemo for 24 weeks. Chemo and DC vaccinations will be given intratumoral and subcutaneous for 4 times prior surgery. During the AC cycles, vaccines will be given on any day between Days 9-12 of Cycles 1 and 3 of AC. Vaccines will be given on any day between Days 11-15 of Cycles 1 and 3 of TCb. Patients will undergo biopsies of their cancer prior to treatment and 1-2 days prior to or on Day 1 of Cycle 4 of AC. After this, patients will have surgery, locoregional radiation therapy to the breast or chest wall and regional lymphatics per standard of care, and will receive 3 boost DC vaccinations subcutaneously, rotating injection sites in the upper arm. The 1st vaccination will occur after the surgery and prior to radiation; 2nd will occur 30 days ± 3 days after radiation; the 3rd will occur 90 days ± 3 days after the 2nd boost.
  Interventions: Biological: LA TNBC: DC vaccine+Preop chemo
- ER+/HER2-BC:DC vaccine+Preop chemo (Experimental): ER+/HER2- BC patients will receive standard preop AC followed by weekly T given for 22 weeks. Chemo and DC vaccinations will be given intratumoral and subcutaneous, for 4 times prior surgery. During the AC cycles, vaccines will be given any day between Days 9-12 of Cycles 1 and 3 of AC. Vaccines will be given on Day 1 during Cycle 2 or Cycle 3 and on Day 1 during either Cycle 8 or Cycle 9 of T. Vaccine will be given after T infusion is completed. Patients will undergo biopsies of their cancer prior to treatment and 1-2 days prior to or on Day 1 of Cycle 4 of AC. Patients will have surgery, locoregional radiation therapy to the breast or chest wall and regional lymphatics per standard of care, and will receive 3 boost DC vaccinations subcutaneously, rotating injection sites in the upper arm. The 1st vaccination will occur after surgery and prior to radiation; the 2nd will occur 30 days ± 3 days after radiation; and the 3rd will occur 90 days ± 3 days after the 2nd boost.
  Interventions: Biological: ER+/HER2-BC:DC vaccine+Preop chemo

INTERVENTIONS:
Biological: LA TNBC: DC vaccine+Preop chemo — LA TNBC patients will receive standard preop AC followed by TCb chemo for 24 weeks. Chemo and DC vaccinations will be given intratumoral and subcutaneous for 4 times prior surgery. During the AC cycles, vaccines will be given on any day between Days 9-12 of Cycles 1 and 3 of AC. Vaccines will be given on any day between Days 11-15 of Cycles 1 and 3 of TCb. Patients will undergo biopsies of their cancer prior to treatment and 1-2 days prior to or on Day 1 of Cycle 4 of AC. After this, patients will have surgery, locoregional radiation therapy to the breast or chest wall and regional lymphatics per standard of care, and will receive 3 boost DC vaccinations subcutaneously, rotating injection sites in the upper arm. The 1st vaccination will occur after the surgery and prior to radiation; 2nd will occur 30 days ± 3 days after radiation; the 3rd will occur 90 days ± 3 days after the 2nd boost.
  Other Names: DC Vaccine - Dendritic Cell Vaccine; Preop chemo: Doxorubicin; Preop chemo: cyclophosphamide; Preop chemo: Paclitaxel; Preop chemo: Carboplatin
  Arms: LA TNBC: DC vaccine+Preop chemo
Biological: ER+/HER2-BC:DC vaccine+Preop chemo — ER+/HER2- BC patients will receive standard preop AC followed by weekly T given for 22 weeks. Chemo and DC vaccinations will be given intratumoral and subcutaneous, for 4 times prior surgery. During the AC cycles, vaccines will be given any day between Days 9-12 of Cycles 1 and 3 of AC. Vaccines will be given on Day 1 during Cycle 2 or Cycle 3 and on Day 1 during either Cycle 8 or Cycle 9 of T. Vaccine will be given after T infusion is completed. Patients will undergo biopsies of their cancer prior to treatment and 1-2 days prior to or on Day 1 of Cycle 4 of AC. Patients will have surgery, locoregional radiation therapy to the breast or chest wall and regional lymphatics per standard of care, and will receive 3 boost DC vaccinations subcutaneously, rotating injection sites in the upper arm. The 1st vaccination will occur after surgery and prior to radiation; the 2nd will occur 30 days ± 3 days after radiation; and the 3rd will occur 90 days ± 3 days after the 2nd boost.
  Other Names: DC Vaccination - Dendritic cell vaccination; Preop chemo - doxorubicin; Preop chemo - cyclophosphamide; Preop chemo - paclitaxel; Preop chemo: Carboplatin
  Arms: ER+/HER2-BC:DC vaccine+Preop chemo

SUMMARY:
The primary objective of this study is to determine the safety and feasibility of combining cyclin B1/WT-1/CEF (antigen)-loaded DC vaccination with preoperative chemotherapy.

The secondary objectives of this trial are to determine pathologic complete response rates; disease-free survival; to assess immune biomarkers of immunity (antigen-specific CD8+ T cell immunity and TH2 T cells) in breast cancer biopsy specimens and blood samples in patients receiving DC vaccinations; and to assess the feasibility of immunizing LA TNBC and ER+/HER2- BC patients with patient-specific tumor antigens.

DETAILED DESCRIPTION:
Recent studies have shown that human breast cancers can be immunogenic, and that enhancing the immune effector function already present may augment the cytotoxic effects of standard therapies.

vaccination remains the most attractive strategy because of its expected inducement of both therapeutic T cell immunity (effector T cells) and protective T cell immunity (tumor-specific memory T cells that can control tumor relapse). Several clinical studies have now demonstrated that immunity against tumor antigens can be enhanced in cancer patients by vaccination with ex vivo-generated tumor antigen-loaded dendritic cells (DCs). This strategy capitalizes on the unique capacity of DCs to prime lymphocytes and to regulate and maintain immune responses.

Our goals are to boost T cell immunity targeted against breast cancer utilizing a tumor antigen-loaded DC vaccine, to enhance chemotherapy effectiveness and decrease tumor metastagenicity, and to decrease the recurrence rates of LA TNBC and ER+/HER2- BC. Patients will be treated with a combination of antigen-loaded DC vaccinations along with standard preoperative chemotherapy, to improve immunogenicity and to increase the pCR rate achieved with standard therapy. The trial will consist of 2 patient cohorts: TNBC and ER+/HER2- BC.

ELIGIBILITY:
- Inclusion Criteria:

A patient will be considered for enrollment in this study if all of the following criteria are met:

1. Female patients ≥18 years of age.
2. Have either:

   1. locally advanced TNBC defined as invasive ductal cancer; ER- tumors with <10% of tumor nuclei immunoreactive; PR- tumors with <10% of tumor nuclei immunoreactive; T3 or T4 disease, regardless of nodal status (T2 disease is eligible if there are positive lymph nodes present by physical exam or imaging evaluation or histological evaluation, OR
   2. High-risk ER+ breast cancer defined as grade 3 invasive ductal or mixed ductal/lobular cancers, or grade 2 with Ki67 ≥20%; node positive as evidenced by physical exam or imaging evaluation or histological evaluation.
3. HER2- negative breast cancer. If HER2-, it is defined as follows:

   1. FISH-negative (FISH ratio <2.0), or
   2. IHC 0-1+, or
   3. IHC 2+ AND FISH-negative (FISH ratio<2.0)
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
5. Adequate hematologic function, defined by:

   1. Absolute neutrophil count (ANC) >1500/mm3
   2. Platelet count ≥100,000/mm3
   3. Hemoglobin >9 g/dL (in the absence of red blood cell transfusion)
6. Adequate liver function, defined by:

   1. AST and ALT ≤2.5 x the upper limit of normal (ULN)
   2. Total bilirubin ≤1.5 x ULN
7. Adequate renal function, defined by:

   a. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance of ≥60 ml/min
8. Patients with previous history of invasive cancers (including breast cancer) are eligible if definitive treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease.
9. Eligible for treatment with paclitaxel, doxorubicin, cyclophosphamide and carboplatine.
10. Patient must be accessible for treatment and follow-up.
11. Patients must be willing to undergo research biopsies to obtain breast cancer tissue for whole exome sequencing and evaluation of tumor immune microenvironment.
12. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

    * Exclusion Criteria:

A patient will be ineligible for inclusion in this study any of the following criteria are met:

1. Evidence of metastatic disease on bone scan and CT scan of chest/abdomen (or PET CT scan). Patients with intrathoracic metastatic adenopathy are eligible.
2. Active infection or unexplained fever >38.5°C during screening.
3. Active infections including viral hepatitis and HIV.
4. Active asthma or other condition requiring steroid therapy.
5. Autoimmune disease including lupus erythematosus or rheumatoid arthritis. Topical or inhaled corticosteroids are allowed.
6. Patients who are currently receiving or who have received previous systemic therapy for breast cancer (eg, chemotherapy, antibody therapy, targeted agents).The use of an LHRH agonist during chemotherapy in premenopausal women who wish to preserve ovarian function is allowed, but is not required.
7. Women who are pregnant or lactating. All patients with reproductive potential must agree to use effective contraception from time of study entry until at least 3 months after the last administration of study drug.
8. Have a NYHA Class III or IV CHF or LVEF <55%. Patients with significant cardiac disease history within 1 year or ventricular arrhythmias requiring medication are also excluded.
9. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as:

   1. severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
   2. uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
   3. liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
10. History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, or that might affect interpretation of the results of this study, or render the patient at high risk for treatment complications.
11. Any other investigational or anti-cancer treatments while participating in this study.
12. Any other cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arm "ER+/HER2- BC: DC vaccine + preop chemo" is not included in these results, as no participants were enrolled in this arm with these hormone receptor criteria.
Groups:
- LA TNBC: DC Vaccine+Preop Chemo: LA TNBC patients will be enrolled to receive DC vaccinations during the 24 weeks of standard preoperative dose-dense doxorubicin/cyclophosphamide (AC) followed by paclitaxel and carboplatin (TCb) chemotherapy.
Period: Overall Study
Arm/Group | LA TNBC: DC Vaccine+Preop Chemo
Started | 10
Completed | 6
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | LA TNBC: DC Vaccine+Preop Chemo
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1
  White | 9
  Not Hispanic or Latino | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety of DC Vaccine Combined With Chemotherapy
Description: Toxicities will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 . This will include all patients (eligible and ineligible) who receive at least 1 inoculation of DC vaccine therapy. This safety population will also be used for the summaries and analysis of all safety parameters (drug exposure, tables of adverse events information, including serious adverse events, etc.).
Time Frame: 4 years
Population: Results are only reported for Arm 1, "LA TNBC: DC vaccine+preop chemo patients". Arm 2, "ER+/HER2- BC: DC vaccine+preop chemo patients" did not enroll any patients with these hormone receptor criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | LA TNBC: DC Vaccine+Preop Chemo
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Pathologic Complete Response Rate
Description: Results are only reported for Arm 1, "LA TNBC: DC vaccine+preop chemo patients". Arm 2 did not enroll any patients.
  The pathologic specimen will be graded per the tumor regression grading schema provided by the University of Texas MD Anderson Cancer Center "Residual Cancer Burden Calculator" at http://www3.mdanderson.org/app/medcalc/index.cfm?pagename=jsconvert3. The following parameters are required from pathologic examination in order to calculate RCB: largest 2 dimensions of residual tumor bed in the breast; entire largest cross-sectional area of residual tumor bed; percentage of the tumor bed area that contains carcinoma; percentage of carcinoma in tumor bed that is in situ; number of positive (metastatic) lymph nodes; largest diameter of largest nodal metastasis. A pathologic complete response is defined as NO pathologic evidence of invasive disease in the breast or axillary lymph nodes. RCB-I (minimal cancer burden); RCB-II (moderate burden); and RCB-III (extensive burden).
Time Frame: 1 year
Population: All eligible patients who have received at least 1 inoculation of DC vaccine therapy will be assessed for pathologic complete response.
Measure: Count of Participants; unit: Participants
Arm/Group | LA TNBC: DC Vaccine+Preop Chemo
Number analyzed (Participants) | 10
Participants
  pathologic complete response (pCR) | 4
  Residual Cancer Burden 1 (RCB1) | 3
  Residual Disease (RD) | 3

3. Secondary Outcome: Disease-free Survival
Description: Results are only reported for Arm 1, "LA TNBC: DC vaccine+preop chemo patients". Arm 2, "ER+/HER2- BC: DC vaccine+preop chemo patients" did not enroll any patients with these hormone receptor criteria.
  Analysis of disease-free survival ("DFS", reported in months) was calculated from the first day of treatment up to 36 months.
Time Frame: 36 months
Population: All eligible patients who have received at least 1 inoculation of DC vaccine therapy.
Measure: Mean (Full Range); unit: months
Arm/Group | LA TNBC: DC Vaccine+Preop Chemo
Number analyzed (Participants) | 10
months | 15.6 [6.5 to 26.32]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Results are only reported for Arm 1, "LA TNBC: DC vaccine+preop chemo patients". Arm 2, "ER+/HER2- BC: DC vaccine+preop chemo patients" did not enroll any patients with these hormone receptor criteria.
  All Grade 2, 3 and 4 adverse events (AEs), Grades 1 and 2 alopecia, and all grades of neutropenia will be recorded in the CRF throughout the trial.
  All AEs will be recorded for up to 30 days following the last study treatment.
Arm/Group | LA TNBC: DC Vaccine+Preop Chemo
All-Cause Mortality (participants affected / at risk) | 4/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LA TNBC: DC Vaccine+Preop Chemo (N=10)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Right atrial thrombosis (Cardiac disorders) | 1
cellulitis of right breast (Skin and subcutaneous tissue disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LA TNBC: DC Vaccine+Preop Chemo (N=10)
Gastroesophageal Reflux (Gastrointestinal disorders) | 4
Hot Flashes (General disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 10
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3
Nodule Left Arm (Skin and subcutaneous tissue disorders) | 1
Tingling (Nervous system disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Fever (General disorders) | 4
Headache (General disorders) | 10
Chills (General disorders) | 1
Mucositis (Gastrointestinal disorders) | 5
Oral Candidiasis (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 8
Gastroenteritis (Gastrointestinal disorders) | 1
Parageusia (Gastrointestinal disorders) | 6
Pruritus (General disorders) | 1
Venous Access Failure (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Right Axilla Pain (Musculoskeletal and connective tissue disorders) | 1
Right breast cellulitis post reconstruction/expanders surgery (Skin and subcutaneous tissue disorders) | 1
Weight loss (General disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Sore Throat (Infections and infestations) | 1
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1
Epistaxis (Vascular disorders) | 2
Sleep Disturbance (General disorders) | 2
Peripheral Neuropathy hands and feet (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Seroma Left Axilla (Musculoskeletal and connective tissue disorders) | 1
Upper Abdomen Pain (Gastrointestinal disorders) | 1
Blurred Vision (General disorders) | 1
Tingling of the Tongue (Nervous system disorders) | 1
Peripheral Neuropathy arms and hands (Nervous system disorders) | 1
Peripheral Neuropathy bilateral feet (Nervous system disorders) | 1
flutter in chest (Cardiac disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 1
UTI (Renal and urinary disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
DVT LLE (Vascular disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2
Intermittent Neuropathy in Toes (Nervous system disorders) | 1
Right breast focal fibrosis with fat necrosis (Skin and subcutaneous tissue disorders) | 1
Numbness of feet (Nervous system disorders) | 1
Fungal infection left great toe (Infections and infestations) | 1
Seroma bilateral breast (Skin and subcutaneous tissue disorders) | 1
Redness Right Breast (Skin and subcutaneous tissue disorders) | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Left big toe brittle nail (Skin and subcutaneous tissue disorders) | 1
Right upper extremity lymphedema (Vascular disorders) | 1
Pain (General disorders) | 1
Chest Pain (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dehydration (General disorders) | 1
Dizziness (General disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Intermittent Neuropathy (Nervous system disorders) | 1
Herpes Genitalis (Infections and infestations) | 1
Anxiety (Psychiatric disorders) | 2
Pain Right Shoulder (General disorders) | 1
Vibrating Apheresis (Investigations) | 2
Tachycardia (Cardiac disorders) | 1
Mouth Sores (Gastrointestinal disorders) | 2
Insect Bite (General disorders) | 1
Mastalgia right breast (Musculoskeletal and connective tissue disorders) | 1
Neuropathy (Nervous system disorders) | 2
Hyperglycemia (Endocrine disorders) | 1
Arthralgias (Musculoskeletal and connective tissue disorders) | 2
Hypovitaminosis (General disorders) | 1
Chemo induced nails bruised (Skin and subcutaneous tissue disorders) | 1
Neuropathy bilateral lower extremity (Nervous system disorders) | 1
Tenderness of lymph nodes in right armpit (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Cardiac disorders) | 1
Joint popping in hands (Musculoskeletal and connective tissue disorders) | 1
Neuropathy in hands and feet (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT02018458/Prot_SAP_000.pdf